CLINICAL TRIAL: NCT06779851
Title: A Phase 1 Investigation of the Safety, Tolerability and Preliminary Antitumor Activity of BPT567, a Multifunctional PD1-IL18 Immunocytokine in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate Safety and Tolerability of BPT567 in Patients With Advanced Solid Tumors
Acronym: SUMMIT-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bright Peak Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BPT567-101
Record Dates: First submitted 2025-01-03; First posted 2025-01-17 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors
Keywords: Solid Tumors

STUDY DESIGN:
Intervention Model Description: Ph1a Dose Escalation followed by and Ph 1b Dose Expansion study including multiple expansion cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a Dose Escalation (Experimental): Study drug BPT567 at multiple dose levels to define MTD or MAD
  Interventions: Drug: BPT567
- Phase 1b Dose Expansion (Experimental): Study drug BPT567 at recommended dose for expansion (RDE) cohorts
  Interventions: Drug: BPT567

INTERVENTIONS:
Drug: BPT567 — Immunocytokine infusion

SUMMARY:
This is a first-in-human Phase Ia/Ib, open-label, multicenter, dose escalation and dose expansion study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and maximum tolerated dose (MTD) or maximum adminstered dose (MAD) of BPT567 in patients with advanced solid tumors, and establish the recommended dose for expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years at the time of signing informed consent form
* Measurable disease per RECIST 1.1
* Histologically- or cytologically-diagnosed, locally advanced unresectable or metastatic solid tumor. Progressed or recurred after previously having received approved standard of care agents that are approved and available in their local geography.
* ECOG Performance status of 0 or 1
* Life expectancy of at least 3 months
* Adequate organ and marrow function
* Contraception during study participation, as applicable

Exclusion Criteria:

* Has received systemic small molecule therapy or radiation therapy within 28 days prior to the first dose.
* Treatment with biologic agents including anti-PD-1 or PD-L1 antibodies for less than 6 weeks or 5 half-lives, whichever is shorter, prior to first dose.
* Received any investigational agent less than 28 days or 5 half-lives, whichever is shorter, prior to the first dose.
* Treatment with another IL-18 therapy.
* Received systemic immunosuppressive agents greater than the equivalent of prednisone 10mg daily within 14 days of the study, though inhaled, intranasal, topical or intra-articular corticosteroids are allowed.
* Certain clinically significant intercurrent disease.
* Primary immune deficiency.
* Active untreated brain or spine metastasis or leptomeningeal metastases.
* Known HIV seroposivitiy, although patients treated for HIV with no detectable viral load for at least 1 month while on a stable regimen of agents are permitted.
* Active hepatitis A or acute or chroming hepatitis B or C infection.
* Received a live virus vaccine within 30 days of enrollment or a COVD vaccine within 14 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT), Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) | Duration of first cycle (28 Days) for each cohort evaluated
  The MTD will be the highest tested dose of BPT567 at which protocol specified number of patients experience DLT or the MAD, highest administered dose in the absence of DLTs
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | Through end of study (up to 2 years)
  Rate of subjects reporting adverse events or serious adverse events including abnormalities in safety laboratory results

SECONDARY OUTCOMES:
Pharmacokinetic parameter - Maximum Concentration (Cmax) | Cycle 1 (Days 1,2, 4, 8, 15 & 22) Cycles 2& 3 (Days 1&15) Cycles 4 & beyond (Day1) End of Treatment (up to 2 years)
  Maximum concentration of BPT567
Pharmacokinetic parameter - Time to Maximumn Concentration (Tmax) | Cycle 1 (Days 1,2, 4, 8, 15 & 22) Cycles 2& 3 (Days 1&15) Cycles 4 & beyond (Day1) End of Treatment (up to 2 years)
  Time to maximum concentration of BPT567
Pharmacokinetic parameter - Terminal Elimination Half-life (T1/2) | Cycle 1 (Days 1,2, 4, 8, 15 & 22) Cycles 2& 3 (Days 1&15) Cycles 4 & beyond (Day1) End of Treatment (up to 2 years)
  Terminal elimination half-life of BPT567
Pharmacokinetic parameter - Area under the plasma concentration curve up to the last quantifiable time-point ((AUC)0-last)) | Cycle 1 (Days 1,2, 4, 8, 15 & 22) Cycles 2& 3 (Days 1&15) Cycles 4 & beyond (Day1) End of Treatment (up to 2 years)
  (AUC)0-last of BPT567
Pharmacokinetic parameter - Area area under the curve from 0 to infinite time (AUC0-inf) | Cycle 1 (Days 1,2, 4, 8, 15 & 22) Cycles 2& 3 (Days 1&15) Cycles 4 & beyond (Day1) End of Treatment (up to 2 years)
  AUC0-inf of BPT567
Anti-drug Antibody (ADA) Response to BPT567 | Predose and postdose at multiple timepoints up to end of treatment (up to 2 years)
  Number of Participants With Anti-drug Antibody (ADA) Response to BPT567
Objective response rate (ORR) | Through study completion up to 2 years
  Per RECIST V1.1
Duration of response (DoR) | Through study completion up to 2 years
  Per RECIST V1.1
Disease Control Rate (DCR) | Through study completion up to 2 years
  Per RECIST V1.1
Progression Free Survival (PFS) | Through study completion up to 2 years
  Per RECIST V1.1

OTHER OUTCOMES:
Evaluate changes in immune cell composition and tumor genome. | Through study completion up to 2 years
  Peripheral blood and/or tumour biopsy specimens may be analysed in an exploratory manner to assess changes in immune cell composition through immunophenotyping and cytokine level measurements.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Start Midwest, Grand Rapids, Michigan
  - Hackensack Meridian John Theurer Cancer Center, Hackensack, New Jersey
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Providence Cancer Institute, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas